CLINICAL TRIAL: NCT04836156
Title: Neoadjuvant Therapy Study Guided by Drug Screening in Vitro Patient-derived Tumor-like Cell Clusters for Human Epidermal Growth Factor Receptor 2 (HER2) Negative Early Breast Cancer Patients
Brief Title: Neoadjuvant Therapy Study Guided by Drug Screening in Vitro for Human Epidermal Growth Factor Receptor 2 (HER2) Negative Early Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUPH10B004
Record Dates: First submitted 2021-03-28; First posted 2021-04-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: HER2-negative Early Breast Cancer
MeSH Terms: interventions — Docetaxel; Carboplatin; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant therapy base on PTC drug screening for triple negative early breast cancer (Experimental): Patients with triple negative subtype will receive neoadjuvant chemotherapy based on PTC drug screening.
  Interventions: Drug: neoadjuvant chemotherapy upon in vitro PTC drug sensitivity screening for triple negative breast cancer
- Neoadjuvant therapy base on PTC drug screening for luminal like early breast cancer (Experimental): Patients with luminal like subtype will receive neoadjuvant chemotherapy based on PTC drug screening.
  Interventions: Drug: neoadjuvant chemotherapy upon in vitro PTC drug sensitivity screening for luminal like breast cancer

INTERVENTIONS:
Drug: neoadjuvant chemotherapy upon in vitro PTC drug sensitivity screening for triple negative breast cancer — The choice of chemotherapy is based on the PTC drug sensitivity results.
  Other Names: docetaxel and carboplatin; docetaxel and epirubicin
  Arms: Neoadjuvant therapy base on PTC drug screening for triple negative early breast cancer
Drug: neoadjuvant chemotherapy upon in vitro PTC drug sensitivity screening for luminal like breast cancer — The choice of chemotherapy is based on the PTC drug sensitivity results.
  Other Names: docetaxel and cyclophosphamide; epirubicin and cyclophosphamide; docetaxel and epirubicin
  Arms: Neoadjuvant therapy base on PTC drug screening for luminal like early breast cancer

SUMMARY:
Neoadjuvant treatment is an important treatment for early breast cancer patients. Patients with triple negative subtype who achieved pCR after neoadjuvant treatment would have longer survival. The neoadjuvant treatment for her2 negative patient was chemotherapy with combined drugs. However, not all patients benefit from chemotherapy but suffer from chemotherapy-related side effects. It was unknown for a patient who could benefit from which drug before chemotherapy. Drug sensitivity screening in vitro was a promising method for choosing chemotherapy. But there was no method could select effective drugs accurately for breast cancer patients until now.

Previously, investigators developed a patient-derived tumor-like cell clusters in vitro culture technology. Feasibility for guiding clinical treatment by drug sensitivity screening based on this technology have been explored by preliminary exploration with a well corresponding. And the results have been published. This study will explore whether drug screening in vitro patient-derived tumor-like cell clusters from breast cancer tissue could be a method for selection of chemotherapy for her2 negative participants.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy for breast cancer could make unresectable breast cancer be resectable and improve breast conservation rate. Patients with triple negative subtype who achieved pCR after neoadjuvant treatment would have longer survival. The neoadjuvant treatment for her2 negative patient was chemotherapy with combined drugs. However, not all patients benefit from chemotherapy but suffer from chemotherapy-related side effects. It was unknown for a patient who could benefit from which drug before chemotherapy. Drug sensitivity screening in vitro was a promising method for choosing chemotherapy. But there was no method could select effective drugs accurately for breast cancer participants until now.

Previously, investigators developed a patient-derived tumor-like cell clusters (PTC) in vitro culture technology. It is a cell cluster including tumor cells, mesenchymal cells and lymphocytes, which simulates the tumor microenvironment in vitro. In the preliminary exploration, investigators included 35 early breast cancer participants, the corresponding between in vitro drug sensitivity screening based on this technology and clinical treatment results was well. The results have been published.

This study will focus on her2 negative early breast cancer participants. 46 participants will be included. All of them will received in vitro drug sensitivity screening upon PTC before neoadjuvant therapy. The choice of chemotherapy drugs is determined based on the PTC drug sensitivity results. If single-agent chemotherapy is effective in vitro, this drug will be the chemotherapy regimen for the corresponding participants.

ELIGIBILITY:
Inclusion Criteria:

* invasive breast cancer
* HER2 negative
* T2 or node positive
* Eastern Cooperative Oncology Group(ECOG) 0-1

Exclusion Criteria:

* stage IV
* inflammatory breast cancer
* Severe chronic disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response(pCR) | up to 24 weeks
  ypT0/is, ypN0

SECONDARY OUTCOMES:
event-free survival (EFS) | 5 years
  The time from random assignment to disease progression, including local progression before surgery; disease recurrence-local, regional, distant, ipsilateral noninvasive, or contralateral (invasive or noninvasive)-or death from any cause
invasive disease-free survival (IDFS) | 5 years
  The time from surgery to the first documented occurrence of an event defined as ipsilateral invasive local recurrence, ipsilateral locoregional invasive recurrence, distant recurrence, contralateral invasive breast cancer, or death from any cause
objective response rate | up to 24 weeks
  complete response and partial response

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China